CLINICAL TRIAL: NCT02336503
Title: A Multicenter, Randomized, Double Blind, Vehicle-Controlled Study to Evaluate the Safety and Effect on Sweat Production of 3 Concentrations of Topically Applied BBI-4000 in Subjects With Axillary Hyperhidrosis
Brief Title: A Safety and Efficacy Study of BBI-4000 in Subjects With Axillary Hyperhidrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Botanix Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BBI-4000-CL-201
Record Dates: First submitted 2015-01-08; First posted 2015-01-13 (Estimated); Results first posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2022-12

CONDITIONS: Hyperhidrosis
MeSH Terms: conditions — Hyperhidrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BBI-4000 Gel, 5% (Experimental): Low concentration of BBI-4000; BBI-4000 Gel, 5%
  Interventions: Drug: BBI-4000 Gel, 5%
- BBI-4000 Gel, 10% (Experimental): Middle concentration of BBI-4000; BBI-4000 Gel, 10%
  Interventions: Drug: BBI-4000 Gel, 10%
- BBI-4000 Gel, 15% (Experimental): High concentration of BBI-4000; BBI-4000 Gel, 15%
  Interventions: Drug: BBI-4000 Gel, 15%
- Vehicle (Placebo Comparator): Vehicle (placebo); BBI-4000 Gel, 0%
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: BBI-4000 Gel, 5% — BBI-4000 Gel, 5%
  Other Names: BBI-4000 Low Dose
  Arms: BBI-4000 Gel, 5%
Drug: BBI-4000 Gel, 10% — BBI-4000 Gel, 10%
  Other Names: BBI-4000 Middle Dose
  Arms: BBI-4000 Gel, 10%
Drug: BBI-4000 Gel, 15% — BBI-4000 Gel, 15%
  Other Names: BBI-4000 High Dose
  Arms: BBI-4000 Gel, 15%
Drug: Vehicle — Placebo, BBI-4000 Gel, 0%
  Other Names: Placebo
  Arms: Vehicle

SUMMARY:
To assess the safety and efficacy of 3 doses of BBI-4000 and vehicle (4 treatment arms), when applied once a day for 4 weeks, for the treatment of axillary hyperhidrosis.

DETAILED DESCRIPTION:
This is a Multicenter, Randomized, Double Blind, Vehicle-Controlled Study to Evaluate the Safety and Efficacy of 3 concentrations of Topically Applied BBI-4000 in Subjects with Axillary Hyperhidrosis.

Participating subjects will apply BBI-4000 once a day for 4 weeks in their axillae. The 4 week treatment period will be followed by a 2 week follow-up period.

Safety will be assessed through collection of vital signs, adverse events, local skin responses, hematology and serum chemistry laboratory testing and ECGs.

Efficacy will be assessed using the Hyperhidrosis Disease Severity Scale (patient reported outcome) and through gravimetrically measured sweat production.

PK blood samples will be taken from study subjects from selected centers.

ELIGIBILITY:
Inclusion Criteria:

* Primary axillary hyperhidrosis of at least 6 months's duration
* Hyperhidrosis disease severity score of 3 or 4 at baseline
* Gravimetric test at baseline indicating at least 50 mg of sweat production at rest in each axilla, in 5 minutes (room temperature)
* Willing to refrain from using any other antiperspirant agent for the duration of the study.
* Females of childbearing potential must agree to use a medically acceptable method of contraception while participating in the study.

Exclusion Criteria:

* Any skin or subcutaneous tissue conditions in the axilla or near the axillary area, other than hyperhidrosis.
* Prior use of any prohibited medication(s) or procedure(s) within the specified timeframe, including:

  1. Botulinum toxin to the axillary area within 1 year of the baseline visit.
  2. Axillary iontophoresis within 12 weeks of baseline visit.
  3. Axillary thermolysis, sympathectomy or surgical procedures of the axillary area at any time in the past.
* Use of systemic and/or topical anticholinergic treatment within 30 days of the baseline visit.
* Subjects with hyperhidrosis symptoms initiated or exacerbated with their menopause.
* Subjects with history of diabetes mellitus, renal impairment, hepatic impairment, thyroid disease, malignancy, glaucoma, intestinal obstructive or motility disease, obstructive uropathy, myasthenia gravis, benign prostatic hyperplasia (BPH), neurological conditions, psychiatric conditions, Sjögren's syndrome, Sicca syndrome, or cardiac abnormalities that may alter normal sweat production or may be exacerbated by the use of anticholinergics.
* Subjects with known hypersensitivity to glycopyrrolate, anticholinergics, or any of the components of the topical formulation.
* Pregnant or lactating women.
* Use of an investigational drug within 30 days prior to the baseline visit.
* Prior treatment with the study drug in a previous trial.
* Any major illness within 30 days before the screening examination.
* Any other condition or laboratory abnormality that, in the judgment of the investigator, would put the subject at unacceptable risk for participation in the study or may interfere with the assessments included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2015-03-10 (Actual); Primary Completion 2015-11-05 (Actual); Study Completion 2015-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Walker, MD PhD, Study Director — Botanix Pharmaceuticals
Locations (12):
- United States (12):
  - Center for Dermatology Clinical Research, Inc., Fremont, California
  - Therapeutics Clinical Research, San Diego, California
  - Center for Clinical and Cosmetic Research, Aventura, Florida
  - International Dermatology Research, Inc., Miami, Florida
  - International Clinical Research, Sanford, Florida
  - Shideler Clinical Research Center, Carmel, Indiana
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Saint Louis University Dermatology, St Louis, Missouri
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - The Center for Skin Research, Houston, Texas
  - Virginia Clinical Research, Inc., Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- BBI-4000 Gel, 5%: BBI-4000 Gel, 5% Applied to both axillae once nightly
- BBI-4000 Gel, 10%: BBI-4000 Gel, 10% Applied to both axillae once nightly
- BBI-4000 Gel, 15%: BBI-4000 Gel, 15% Applied to both axillae once nightly
- Vehicle: Vehicle (placebo) applied to both axillae nightly
Period: Overall Study
Arm/Group | BBI-4000 Gel, 5% | BBI-4000 Gel, 10% | BBI-4000 Gel, 15% | Vehicle
Started | 47 | 48 | 48 | 46
Completed | 45 | 45 | 47 | 40
Not Completed | 2 | 3 | 1 | 6
Not completed — Lost to Follow-up | 0 | 3 | 0 | 2
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 4
Not completed — Adverse Event | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Population (N=189) was defined as all randomized subjects
Groups:
- BBI-4000 Dose 1: Low concentration of BBI-4000
  BBI-4000 Low Concentration: BBI-4000 Low Dose
- BBI-4000 Dose 2: Middle concentration of BBI-4000
  BBI-4000 Middle Concentration: BBI-4000 Middle Dose
- BBI-4000 Dose 3: High concentration of BBI-4000
  BBI-4000 High Concentration: BBI-4000 High Dose
- Vehicle: Vehicle (placebo)
  Placebo: Vehicle
- Total: Total of all reporting groups
Arm/Group | BBI-4000 Dose 1 | BBI-4000 Dose 2 | BBI-4000 Dose 3 | Vehicle | Total
Number analyzed (Participants) | 47 | 48 | 48 | 46 | 189
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.6 (10.34) | 33.4 (10.61) | 35.5 (11.64) | 32.4 (8.23) | 33.5 (10.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 25 | 27 | 27 | 103
  Male | 23 | 23 | 21 | 19 | 86
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 12 | 11 | 13 | 49
  Not Hispanic or Latino | 34 | 36 | 37 | 33 | 140
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 1 | 3
  Asian | 0 | 0 | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 11 | 13 | 9 | 11 | 44
  White | 35 | 34 | 35 | 32 | 136
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Achieving at Least 2-point Decrease in Hyperhidrosis Disease Severity Scale (HDSS) From Baseline to Week 4
Description: Severity is scored with increasing scale, scores 1-4 where minimal severity is scored: 1=My sweating is never noticeable and never interferes with my daily activities and most severe score is: 4=My sweating is intolerable and always interferes with my daily activities
Time Frame: Baseline through Week 4 (Day 29)
Population: Randomized subjects with reported scores on Baseline and Day 29 (week 4), Count of participants includes number of participants who did not report at-least a 2-point decrease in score (NO) and number of participants who did report at-least a 2-point decrease in score (YES); proportions were calculated as percentages = (# of participants/total # of participants that provided baseline and day 29 HDSS scores) x 100%
Measure: Count of Participants; unit: Participants
Groups:
- BBI-4000 Gel, 5%: Low concentration of BBI-4000
  BBI-4000 Gel, 5% Applied to both axillae once nightly
- BBI-4000 Gel, 10%: Middle concentration of BBI-4000
  BBI-4000 Gel, 10% Applied to both axillae once nightly
- BBI-4000 Gel, 15%: High concentration of BBI-4000
  BBI-4000 Gel, 15% Applied to both axillae once nightly
Arm/Group | BBI-4000 Gel, 5% | BBI-4000 Gel, 10% | BBI-4000 Gel, 15% | Vehicle
Number analyzed (Participants) | 47 | 47 | 47 | 41
Participants
  No | 35 | 37 | 29 | 36
  Yes | 12 | 10 | 18 | 5

2. Secondary Outcome: Proportion of Subjects Achieving at Least 1-point Improvement in Hyperhidrosis Disease Severity Scale (HDSS) From Baseline to Week 4
Description: as for outcome 1
Time Frame: Baseline through Week 4 (Day 29)
Population: Randomized subjects with reported scores on Baseline and Day 29 (week 4), Count of participants includes number of participants who did not report at-least a 1-point decrease in score (NO) and number of participants who did report at-least a 1-point decrease in score (YES); proportions were calculated as percentages = (# of participants YES or NO/total # of participants that provided baseline and day 29 HDSS scores) x 100%
Measure: Count of Participants; unit: Participants
Arm/Group | BBI-4000 Gel, 5% | BBI-4000 Gel, 10% | BBI-4000 Gel, 15% | Vehicle
Number analyzed (Participants) | 47 | 47 | 47 | 41
Participants
  No | 25 | 26 | 13 | 23
  Yes | 22 | 21 | 34 | 18

3. Secondary Outcome: Absolute Change in Gravimetrically Measured Sweat Production From Baseline to Week 4 (Day 29)
Description: Sweat production unit of measure was weight-based (mg); absolute change was calculated by adding the left and right axillae sweat weights and calculating absolute change by subtracting day 29 from baseline sweat weights
Time Frame: Baseline through Week 4 (Day 29)
Population: Randomized participants that provided samples for gravimetric measured sweat production: baseline and day 29
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | BBI-4000 Gel, 5% | BBI-4000 Gel, 10% | BBI-4000 Gel, 15% | Vehicle
Number analyzed (Participants) | 47 | 47 | 47 | 41
mg | -183.1 (370.85) | -56.4 (277.81) | -171.9 (344.54) | -172.9 (315.89)

4. Secondary Outcome: Percent Change in Gravimetrically Measured Sweat Production From Baseline to Week 4
Description: Randomized participants that provided samples for gravimetric sweat measures, baseline and day 29; Percent Change was calculated by dividing absolute change by baseline gravimetric measurement x 100%
Time Frame: Baseline through Week 4 (Day 29)
Population: Randomized participants that provided samples for gravimetric sweat measures, baseline and day 29;
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | BBI-4000 Gel, 5% | BBI-4000 Gel, 10% | BBI-4000 Gel, 15% | Vehicle
Number analyzed (Participants) | 47 | 47 | 47 | 41
percentage of change | -31.9 (84.95) | -15.7 (115.03) | -35.7 (65.48) | -41.7 (40.73)

ADVERSE EVENTS:
Time Frame: Adverse events were assessed following a participant's consent to participate, while receiving approximately one month of investigational treatment (Baseline Visit and Visit Day 29), and subsequently two weeks following completion of investigational treatment (Day 42).
Description: Adverse event definitions followed clinicaltrials.gov guidance
Groups:
- BBI-4000 Gel, 5%: BBI-4000 Gel, 5%, administered to each axillae nightly
- BBI-4000 Gel, 10%: BBI-4000 Gel, 10%, administered to each axillae nightly
- BBI-4000 Gel, 15%: BBI-4000 Gel, 15%, administered to each axillae nightly
- Vehicle: BBI-4000 Gel, 0% (Placebo)
Arm/Group | BBI-4000 Gel, 5% | BBI-4000 Gel, 10% | BBI-4000 Gel, 15% | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/48 | 0/48 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/48 | 0/48 | 0/46
Other Adverse Events (participants affected / at risk) | 8/47 | 12/48 | 14/48 | 6/46
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BBI-4000 Gel, 5% (N=47) | BBI-4000 Gel, 10% (N=48) | BBI-4000 Gel, 15% (N=48) | Vehicle (N=46)
Dry Eye (Eye disorders) | 0 | 1 | 0 | 0
Vision Blurred (Eye disorders) | 2 | 2 | 3 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Dry Mouth (Gastrointestinal disorders) | 2 | 2 | 4 | 0
Eructation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Lip Dry (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Tooth Ache (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Application Site Dermatitis (General disorders) | 2 | 0 | 1 | 0
Application Site Dryness (General disorders) | 0 | 0 | 1 | 0
Application Site Erythema (General disorders) | 0 | 0 | 1 | 0
Application Site Pain (General disorders) | 2 | 2 | 1 | 0
Application Site Pruritus (General disorders) | 2 | 1 | 0 | 0
Application Site Rash (General disorders) | 0 | 2 | 0 | 0
Application Site Swelling (General disorders) | 0 | 0 | 1 | 0
Application Site Folliculitis (Infections and infestations) | 0 | 1 | 1 | 0
Bacterial Vaginosis (Infections and infestations) | 0 | 0 | 0 | 1
Dermatitis Infected (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Herpes Simplex (Infections and infestations) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 2
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 2
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0
Joint Dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tooth Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Crystal Urine Present (Investigations) | 1 | 0 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary Hesitation (Renal and urinary disorders) | 0 | 0 | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Agreement terms prioritized a multi-center publication at the study end. Should such a publication not be completed, an investigator right to individually publish results of his/her study (limited to his/her site data) was included, if for purely scientific or educational purposes; not for any commercial purposes. PI(s) were to submit draft materials to the Sponsor 60 days prior to Investigator release of individual abstract or manuscript. Additional disclosure restrictions and terms applied .